CLINICAL TRIAL: NCT02255071
Title: The Efficacy of Neiguan (P6 Point) Acupressure in Patients With Gastroesophageal Reflux Disease (GERD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CMUH103-REC2-058
Record Dates: First submitted 2014-09-30; First posted 2014-10-02 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: GERD; Neiguan; Acupressure; P6
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupressure (Experimental): Patients will band a acupressure wristband over Neiguan (P6 point) and acupressure for seven days.
  Interventions: Device: Acupressure wristband
- Sham-Acupressure (Sham Comparator): Patients will band a sham wristband over wrist but no acupressure for seven days.
  Interventions: Device: Sham wristband

INTERVENTIONS:
Device: Acupressure wristband — A acupressure wristband over Neiguan (P6 point) and acupressure for seven days.
  Arms: Acupressure
Device: Sham wristband — A wristband over wrist but no acupressure for seven days.
  Arms: Sham-Acupressure

SUMMARY:
In recent years, there is an increasing trend in the number of patients with Gastroesophageal reflux disease (GERD). The poor response to medicine was noticed in patients with non-erosive reflux disease. According to the theory of traditional Chinese medicine, acupuncture Neiguan (P6 point) could improve the uncomfortable symptoms of the chest and upper abdomen. Therefore, the aim of this study is to investigate the clinical efficacy of Neiguan (P6 point) acupressure in patients with GERD.

DETAILED DESCRIPTION:
In recent years, there is an increasing trend in the number of patients with GERD. GERD mainly related to the reflux of stomach content induced by the dysfunction of lower esophageal sphincter. The common symptoms of GERD are heartburn, acid regurgitation, and chest pain. The methods to treat GERD are changes of lifestyle, pharmacotherapy, antireflux surgery and endoscopy. However, the poor response to medicine was still noticed in patients with non-erosive reflux disease. And long-term use of medicine will result in many side effects including infectious, abdominal pain, diarrhea and osteoporosis. According to the theory of traditional Chinese medicine, acupuncture Neiguan (P6 point) could improve the uncomfortable symptoms of the chest and upper abdomen. Therefore, the aim of this study is to investigate the clinical efficacy of Neiguan (P6 point) acupressure in patients with GERD. 64 patients with GERD were randomly divided into two groups：the acupressure and control. In the acupressure group, in addition to receiving standard treatment, patients will band a hand ring over Neiguan (P6 point) and acupressure for seven days. In the control group, in addition to receiving standard treatment, patients will band a hand ring but no acupressure for seven days. Data was collected by self-recorded symptoms before and after the intervention, according to the Reflux disease questionnaire(RDQ) and the World Health Organization Quality of Life Questionnaire Taiwan condensed version. Data was analyzed by Student's t-tests, Paired Student's t-test, Chi-square, and Fisher exact tests for quantitative and qualitative variables. We anticipate the treatment of Neiguan (P6 point) acupressure will reduce the symptoms of gastroesophageal reflux and improve the quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Age of 20-60 years
3. Suffered from heartburn with or without acid regurgitation

Exclusion Criteria:

1. Suffered from peptic ulcer, gallstones, cancer, and Barrett's esophagus
2. previously underwent the esophagus, stomach or duodenum surgery
3. Lactating women or pregnant women
4. patients with severe cardiovascular disease

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-08 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Reflux disease questionnaire(RDQ) | 7 days
  RDQ to assess the severity of GERD for each patient over the past 7 days before study and after banding a wristband for 7days.

SECONDARY OUTCOMES:
World Health Organization Quality of Life Questionnaire Taiwan condensed version(WHOQOL-REF) | 7 days
  WHOQOL-REF(Taiwan version) to assess the Quality of Life for each patient before study and after banding a wristband for 7days.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Ti Hsu, MD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan